CLINICAL TRIAL: NCT06258122
Title: Evolution Over 15 Years (2008-2023) of the Clinical, Immuno-virological and Aging Trajectory of Patients Living With HIV
Brief Title: Evolution of the Clinical, Immuno-virological and Aging Trajectory of Patients Living With HIV
Acronym: TEMPO2
Status: Recruiting | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 17
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Main objective is:

* To characterize the evolution of the immuno-virological profile of circulating blood cells and immune aging in patients who had participated to TEMPO-1 in 2007-2008
* To evaluate the role of immune aging and inflammatory profile in the occurrence of comorbidities in HIV-infected individuals over a 15-year period

The alterations that affect the innate and adaptive immune cell compartments in HIV-infected patients are reminiscent of the process of immune aging, characteristic of old age. These alterations, the presumed cause of which is the chronic systemic immune activation established in patients, contribute to the depletion of lymphoid resources which probably leads to the decline of immune competence with the progression of HIV disease.

The comparison between HIV-1-infected patients and uninfected older adults goes beyond the mere appearance of immunosenescence and extends to the deterioration of a number of physiological functions linked to inflammation and to systemic aging.

By inducing persistent and lasting immune activation, HIV-1 infection is now considered a model of accelerated immunosenescence and systemic aging. During this process, the immune system quickly becomes exhausted, because the source of its exhaustion (i.e. HIV) cannot be eliminated.

To determine which factors may contribute to immunosenescence in HIV-1 infection, we propose an extensive immune and virological evaluation in patients who participated in a cross-sectional assessment of immune functions and TEMPO-1 viral reservoirs after 15 years of evolution in order to determine their immune and viral trajectories, to compare these trajectories with the major clinical events and the comorbidities occurring in them.

DETAILED DESCRIPTION:
Growing old with HIV has become a reality thanks to major advances in antiretroviral therapy. Nearly 40 years after the discovery of the AIDS virus, there are more and more seniors living with HIV. Currently, the median age of HIV-positive people in France is 49 years old. 50% of HIV-positive people are over 50 years old (compared to 8.5% in 1993, 28% in 2010) and 16% over 60 years old. As for discoveries of seropositivity, 20% are in people over 50 years old. According to data from the Dutch ATHENA cohort, the proportion of HIV-infected people aged 50 and over is expected to increase to 73% in 2030.

Thus, if HIV infection has become a chronic disease, with lower mortality Investigator observe a consequent increase in age-related non-infectious comorbidities. Total healthy life expectancy remains reduced among PLHIV compared to uninfected people of the same age, and more than 50% of deaths are due to non-AIDS comorbidities. This polypathology occurs more frequently and at a younger age than in the general population, and notably combines cancers, risk factors and cardiovascular diseases, neurocognitive, bone diseases and chronic renal insufficiency. In 2030, it is estimated that 84% of PLHIV will have at least one of these comorbidities (vs. 29% in 2010), and that 28% will have at least 3, mainly cardiovascular. Some of these comorbidities are linked to the long-term use of ARVs (reverse transcriptase inhibitors, protease inhibitors, integrase inhibitors) leading in particular to metabolic toxicities (dyslipidemia, insulin resistance), renal, bone, endothelial and mitochondrial. However, these toxicities have decreased over time and with pharmacological progress.

n addition to individual or environmental factors such as smoking, a sedentary lifestyle, and classic cardiovascular risk factors, HIV seems to contribute to an acceleration of aging.

The finding of an increased prevalence of non-HIV-related comorbidities such as cardiovascular disease, cancer, renal failure, liver disease, osteopenia and osteoporosis, as well as neurocognitive impairments is reminiscent of classic complications among elderly people with a biological profile marked by inflammation.

Another point in common between PLHIV and the elderly is their prolonged exposure to medications, often constituting polypharmacy.

Thus, antiretroviral molecules, taken by patients for decades for the majority of them, have unfortunately been responsible for various toxicities. First generation ARVs caused cellular disorders with mitochondrial damage for NRTIs such as zidovudine, didanosine or stavudine, metabolic disorders with protease inhibitors. However, the most recent class of molecules, INIs, is not free from toxicities. Indeed, several studies have shown abnormal weight gain with a risk of diabetes and more recently hypertension.

The biological hallmarks of aging are now better understood and include stem cell exhaustion, genomic instability, telomere attrition, impaired intercellular communication, epigenetic alterations, loss of proteostasis, mitochondrial dysfunction and cellular senescence.

Immunologically, aging is associated with a decline in the competence of the immune system called immunosenescence. It is characterized by several features that affect the adaptive and innate immune compartment, as well as the hematopoietic compartment. It is also associated with a high level of secretion of pro-inflammatory cytokines at baseline, called "inflammation", leading to a decreased ability to mount an effective immune response to antigens. Investigators classically describe:

* A decrease in the number of naive T lymphocytes (LT), secondary to thymic involution
* An accumulation of memory cells and a restriction of the antigen receptor repertoire. This is notably determined by the involution of the thymus and the persistence of infectious agents such as cytomegalovirus,
* Shortening of telomeres
* Changes in the gene expression profile within T lymphocyte subpopulations affecting both surface markers and chemokine/cytokine receptors, effector molecules or transcription players.
* A low-grade chronic systemic inflammatory condition called "inflamm-aging". It is characterized by the increased production of proinflammatory cytokines such as IL-1, IL-6, "tumor necrosis factor alpha" (TNF-α) as well as the production of C-reactive protein (CRP). The level of this proinflammatory state is associated with a worse prognosis in elderly patients: increased morbidity and mortality, sarcopenia and frailty.

These global immune changes observed with age contribute in particular to morbidity and mortality linked to infections (in particular via a reduction in the vaccine response) and cancers.

In 2007/2008, with the aim of describing and understanding the different viral and immune phenomena in treated or untreated PLHIV, we carried out a cross-sectional observational study on 240 patients carrying HIV-1.

The TEMPO study included a similar assessment of immune performance in an age- and sex-matched control population. This TEMPO study allowed us to establish the following conclusions:

* massive depletion of CD4+ T cells occurs during HIV-1 infection, such that maintenance of adequate levels of CD4+ T cells depends primarily on the ability to replenish depleted lymphocytes, i.e. - say lymphopoiesis.
* Marked deficiency of primary lymphoid immune resources is seen with failure to maintain adequate lymphocyte numbers.
* Systemic immune activation has emerged as a major correlate of impaired lymphopoiesis, which can be partially reversed by prolonged antiretroviral therapy.

Importantly, disease progression despite elite control of HIV replication or virologic success on antiretroviral therapy has been associated with persistent damage to the lymphopoietic system or exhaustion of lymphopoiesis.

These results highlight the importance of primary hematopoietic resources in HIV pathogenesis and response to antiretroviral therapy.

TEMPO-2 is a cross-sectional study of PLHIV which will evaluate in depth the immuno-virological status of 100 patients studied in the same way 15 years ago (TEMPO-1). The complete history of clinical and biological events will be analyzed over their 15 years of follow-up in the same hospital.

The study includes two groups: one comprising HIV-infected patients (100 PLHIV) and the second comprising subjects not infected with HIV. Both groups participated in the initial study (TEMPO-1) conducted 15 years ago, with an in-depth assessment of immune and virological status.

The immune aging index of this HIV population will be compared to that of a control population of non-HIV subjects who both participated in TEMPO-1 in 2007/2008.

Investigator will focus on the dynamics of immune resources, particularly on hematopoietic progenitors. This approach will allow us to follow the biological trajectory of relevant immune factors and assess how these variables evolve over time between the two time points.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation to the TEMPO-1 study
* 18 years of age or older
* HIV-infected individuals and non-HIV infected control group
* Be affiliated or beneficiary of a social security scheme
* Have signed the consent form.

Exclusion Criteria:

* Subject under " sauvegarde de justice " (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals and non-HIV infected control group
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
measure of number of participants with the frequency of circulating leukocyte cells | one year
  Assessment of 32 biomarkers by Cytek Aurora cytometry to identify more than 15 populations of immune cells
measureof number of participants with the number of hematopoietic stem cells in peripheral blood and their ability to develop a myeloid or lymphoid lineage in culture | one year
  Assessment by culture

SECONDARY OUTCOMES:
measure of number of participants with cytokines and chemokines, being associated with the appearance of comorbidities | one year
  Assessment by ultra-sensitive manner (Luminex and Quantérix technique)
Measure of number of participants with Microbial translocation markers | one year
  Assessment by Elisa technique
Measure of number of participants with the HIV viral reservoir (DNA) | one year
  Assessment by HIV DNA viral load (quantitative analysis) and by Sequencing of HIV in its DNA form (qualitative analysis: presence of resistance mutations, stop codons, insertions/deletions)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France